CLINICAL TRIAL: NCT07272135
Title: A Double-blind, Placebo-controlled, Ascending-dose Study to Assess the Safety, Tolerability and Efficacy of TR4, a Selective β2-adrenoceptor (β2-AR) Antagonist, in Patients With Mild-to-moderate Asthma
Brief Title: Selective β2-AR Antagonism in Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T-030
Record Dates: First submitted 2022-11-21; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The Phase 1 trial is randomised, double-blind, placebo-controlled, and ascending-dose in design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR4 (Experimental): After a run-in period of 2 weeks, 9 patients will be randomly assigned to the TR4 treatment arm. These 9 patients will take incremental doses of 2.5, 5, 10, and 20 mg of TR4, each dose three times daily for 7 days, and then 40 mg three times daily for 21 days, over a total period of 7 weeks.
  Interventions: Drug: TR4
- Placebo (Placebo Comparator): Three patients will take matching placebo capsules in a similar manner to TR4.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TR4 — TR4 is a selective beta-2-adrenoceptor antagonist. TR4 will be weighed into opaque capsules and released for individual patients, in accordance with good manufacturing practice (GMP).
  Arms: TR4
Other: Placebo — Placebo capsules will contain start in opaque capsules.
  Arms: Placebo

SUMMARY:
The objectives are to assess the safety, tolerability and effect on the airways of TR4 in patients with mild-to-moderate asthma. The Phase 1 trial is randomised, double-blind, placebo-controlled, and ascending-dose in design.

DETAILED DESCRIPTION:
After a run-in period of 2 weeks, 12 eligible patients will be randomised to treatment with either TR4 or placebo. Nine patients will take incremental doses of 2.5, 5, 10 and 20 mg of TR4 capsules, each dose three times daily for 7 days, and then 40 mg three times daily for 21 days, over a total period of 7 weeks. Three patients will take matching placebo capsules in a similar manner.

The number of visits and the types are as follows. There will be a maximum of 10 visits to Hammersmith Medicines Research (HMR) for those subjects who complete the whole study according to the protocol. Visit 1 is an out-patient visit for informed consent and screening. Visit 2 is a short out-patient visit at the start of a 2-week run-in period for those subjects who pass screening. After the run-in period, patients who are still eligible will be given a schedule for 8 further visits (Visits 3-10). Participants will stay on the ward for 2 nights during 5 of those visits (Visits 3-7), and for 1 night during Visit 10. Visits 8 and 9 are short out-patient visits. The study will take each subject ~10 weeks to complete. For purposes of data collection and management the study is divided into one session for screening, a run-in period and 5 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Minimum 21 years old
* History of mild-to-moderate asthma for at least 6 months and controlled by an inhaled SABA, as required
* Otherwise healthy
* Ideally have participated in previous asthma studies
* No corticosteroid for whatever reason within 8 weeks of the start of dosing
* No other prescription medicine within 28 days (apart from a short acting beta-agonist (SABA) or contraceptives in women)
* No over-the-counter medicine within 7 days (apart from acetaminophen) before the start of dosing
* Negative screen for drugs of abuse; forced expiratory volume in 1 second (FEV1) more than or equal to 70% predicted
* Fractional exhaled nitric oxide (FeNO) more than or equal to 35 ppb
* 15% fall in FEV1 after inhaled mannitol (PD15)
* Non-smoker or past smoker (<5 pack years)
* Substitution of subject's SABA inhaler with an anti-cholinergic inhaler, ipratropium bromide, for use as a reliever or rescue medication during a run-in period and during dosing with TR4 or placebo.

Exclusion Criteria:

* Positive test for hepatitis B & C or HIV
* Drug or alcohol abuse
* Airway infection or asthma exacerbation in the last 4 weeks
* Current seasonal asthma
* History of emergency treatment of asthma
* Loss of more than 400 mL blood, or participation in other clinical trials of unlicensed medicines within the previous 3 months
* Consumption of grapefruit or herbal remedies within the past 7 days
* Objection by the subject's general practitioner (GP)
* Subjects who are sexually active and not using reliable contraception
* Women who are lactating, pregnant or plan to become pregnant during the study period
* Positive polymerase chain reaction (PCR) test for SARS-CoV-2 virus
* Subjects who have not received both doses of a COVID-19 vaccine.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Mannitol (PD15) | Baseline (day -1) of treatment periods 1 to 5.
  The dose of mannitol causing a 15% fall in FEV1
Mannitol (PD15) | Day 21 of treatment period 5.
  The dose of mannitol causing a 15% fall in FEV1
Spirometry (FEV1) | Day 1 of treatment periods 1 to 5.
  Lung function test: The forced expiratory volume in 1 second (FEV1).
Spirometry (FEV1) | Day 2 of treatment periods 1 to 5.
  Lung function test: The forced expiratory volume in 1 second (FEV1).
Spirometry (FEV1) | Day 21 of treatment period 5.
  Lung function test: The forced expiratory volume in 1 second (FEV1).
Spirometry (FVC) | Day 1 of treatment periods 1 to 5
  Lung function test: forced vital capacity (FVC)
Spirometry (FVC) | Day 2 of treatment periods 1 to 5
  Lung function test: forced vital capacity (FVC).
Spirometry (FVC) | Day 21 of treatment period 5
  Lung function test: forced vital capacity (FVC).
Spirometry (FEF 25-75) | Day 1 of treatment periods 1 to 5
  Lung function test: forced mid-expiratory flow (FEF 25-75) is the mean forced expiratory flow during the middle half of the FVC.
Spirometry (FEF 25-75) | Day 2 of treatment periods 1 to 5
  Lung function test: the forced mid-expiratory flow (FEF 25-75) is the mean forced expiratory flow during the middle half of the FVC.
Spirometry (FEF 25-75) | Day 21 of treatment period 5.
  Lung function test: forced mid-expiratory flow (FEF 25-75) is the mean forced expiratory flow during the middle half of the FVC
Spirometry (FEV1/FVC) | Day 1 of treatment periods 1 to 5.
  Lung function test: FEV1 as a percentage of FVC (FEV1/FVC).
Spirometry (FEV1/FVC) | Day 2 of treatment periods 1 to 5.
  Lung function test: FEV1 as a percentage of FVC (FEV1/FVC).
Spirometry (FEV1/FVC) | Day 21 of treatment period 5.
  Lung function test: FEV1 as a percentage of FVC (FEV1/FVC).
Impulse oscillometry (IOS) (R5, R5-R20) | Change between baseline (day -1) and day 1 of treatment periods 1 to 5.
  Lung function test: A Jaeger impulse oscillometer will be used to obtain measurements according to the investigators standard operating procedure (SOP) and a published algorithm. The following settings will be used for IOS: oscillometric pressure impulses will be superimposed onto the tidal breathing of the subject, for about 30 s, with a pulse sequence of 5 per second and a frequency spectrum between 5 and 35 Hz. Resistance (R) at 5-20 Hz (R5 and R5-R20) during normal tidal breathing will be measured.
IOS (R5, R5-R20) | Day 21 of treatment period 5.
  Lung function test: A Jaeger impulse oscillometer will be used to obtain measurements according to the investigators SOP and a published algorithm. The following settings will be used for IOS: oscillometric pressure impulses will be superimposed onto the tidal breathing of the subject, for about 30 s, with a pulse sequence of 5 per second and a frequency spectrum between 5 and 35 Hz. Resistance (R) at 5-20 Hz (R5 and R5-R20) during normal tidal breathing will be measured.
IOS (AX) | Change between baseline (day -1) and day 1 of treatment periods 1 to 5.
  Lung function test: A Jaeger impulse oscillometer will be used to obtain measurements according to the investigators SOP and a published algorithm. The following settings will be used for IOS: oscillometric pressure impulses will be superimposed onto the tidal breathing of the subject, for about 30 s, with a pulse sequence of 5 per second and a frequency spectrum between 5 and 35 Hz. Reactance (X) at 5-20 Hz (AX) during normal tidal breathing will be measured.
IOS (AX) | Day 21 of treatment period 5.
  Lung function test: A Jaeger impulse oscillometer will be used to obtain measurements according to the investigators SOP and a published algorithm. The following settings will be used for IOS: oscillometric pressure impulses will be superimposed onto the tidal breathing of the subject, for about 30 s, with a pulse sequence of 5 per second and a frequency spectrum between 5 and 35 Hz. Reactance (X) at 5-20 Hz (AX) during normal tidal breathing will be measured.
Airway nitric oxide (FeNO) | Change between baseline (day -1) and day 1 of treatment periods 1 to 5.
  FeNO will be measured using the NIOX Viro handheld electronic device.
Airway nitric oxide (FeNO) | Day 21 of treatment period 5.
  FeNO will be measured using the NIOX Viro handheld electronic device.
Blood eosinophils | Day -1 of treatment periods 1 to 5.
  Blood eosinophils concentration will be used as an inflammatory marker.
Blood eosinophils | Day 21 of treatment period 5.
  Blood eosinophils concentration will be used as an inflammatory marker.

SECONDARY OUTCOMES:
Vital signs (safety): Blood pressure | Day 1 and 2 of treatment periods 1 to 5. Day 21 and 22 of treatment periods 3 to 5.
  Vital signs are assessed to determine safety and tolerability of treatment.
Vital signs (safety): Heart rate | Day 1 and 2 of treatment periods 1 to 5. Day 21 and 22 of treatment periods 3 to 5.
  Vital signs are assessed to determine safety and tolerability of treatment.
Vital signs (safety): Respiratory rate | Day 1 and 2 of treatment periods 1 to 5. Day 21 and 22 of treatment periods 3 to 5.
  Vital signs are assessed to determine safety and tolerability of treatment.
Vital signs (safety): Oral temperature | Day 1 and 2 of treatment periods 1 to 5. Day 21 and 22 of treatment periods 3 to 5.
  Vital signs are assessed to determine safety and tolerability of treatment.
Safety tests of blood and urine | Day 1 of treatment periods 1 to 5 and day 22 of treatment periods 3 to 5.
  Blood and urine for safety tests will be collected before dosing. Blood will be taken for haematology (2 mL in EDTA), and biochemistry and serology (2 x 3.5 mL).
12-lead ECG: Ventricular rate (safety) | Day 1 of treatment periods 1 to 5 and day 22 of treatment periods 3 to 5.
  12-lead ECG will be taken to assess safety and tolerability of treatment. Ventricular rate will be assessed.
12-lead ECG: PR interval (safety) | Day 1 of treatment periods 1 to 5 and day 22 of treatment periods 3 to 5.
  12-lead ECG will be taken to assess safety and tolerability of treatment. The PR interval is the time from the onset of the P wave to the start of the QRS complex.
12-lead ECG: QRS (safety) | Day 1 of treatment periods 1 to 5 and day 22 of treatment periods 3 to 5.
  12-lead ECG will be taken to assess safety and tolerability of treatment. The QRS complex is the combination of the Q, R and S waves.
12-lead ECG: QT interval (safety) | Day 1 of treatment periods 1 to 5 and day 22 of treatment periods 3 to 5.
  12-lead ECG will be taken to assess safety and tolerability of treatment. Corrected QT interval using the Frederica formula (QTcF).
ECG telemetry: Ventricular rate (safety) | Day 1 of treatment periods 1 to 5.
  The ECG will be monitored continuously from 30 min before until 24h after dosing, using a SpaceLabs system.
ECG telemetry: PR interval (safety) | Day 1 of treatment periods 1 to 5.
  The ECG will be monitored continuously from 30 min before until 24h after dosing, using a SpaceLabs system.
ECG telemetry: QRS (safety) | Day 1 of treatment periods 1 to 5.
  The ECG will be monitored continuously from 30 min before until 24h after dosing, using a SpaceLabs system.
ECG telemetry: QT interval (safety) | Day 1 of treatment periods 1 to 5.
  The ECG will be monitored continuously from 30 min before until 24h after dosing, using a SpaceLabs system.
Peak expiratory flow rate (PEFR) | Day -1 to 6 for treatment periods 1 and 2. Day -1 to 7 and day 8 and 16 of treatment periods 3 to 5. Day 21 of treatment period 5.
  Subjects will be given a PEFR meter. A drop of 20% of a subject's normal PEFR is considered in the normal range.
FEV1 (safety) | Day -1 of treatment periods 1 to 5.
  Forced expiratory volume in 1 second.
Pulse oximetry | Day 1 and 2 of treatment periods 1 to 5. Day 21 of treatment periods 3 to 5.
  Pulse oximetry is a non-invasive method for monitoring the saturation of oxygen in the peripheral blood, which will be measured using the SpaceLabs Patients Care Monitoring System (PCMS) and a standard HMR SOP.

OTHER OUTCOMES:
Plasma TR4 and metabolite concentration | Blood samples (4 mL) will be taken on day 1 of treatment periods 1 to 5.
  Plasma concentrations of TR4 and metabolites will be listed and summarised by treatment, using descriptive statistics. Individual pharamcokinetic (PK) parameters will be calculated.
Plasma annexin-A1 | Blood samples (5 mL) will be taken on day -1 of treatment periods 1 to 5 and day 21 of treatment period 5.
  Annexin-A1 is a global anti-inflammatory protein and its receptor levels are known to be modulated in asthmatics. The investigators are using it as an inflammatory biomarker and will measure concentration in plasma using a validated ELISA method.
Lymphocyte beta-2-adrenoceptor density | Blood samples (8 mL) will be taken on day -1 of treatment periods 1 to 5 and day 21 of treatment period 5.
  Flow-cytometry assay used to measure cell-surface density of beta-2-adrenoceptor on lymphocyte subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Denisa Wilkes, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No